CLINICAL TRIAL: NCT03553706
Title: Interference Indicators of Growth, Nutritional Status and Comorbid Malformations of Newborns With Down Syndrome (DS)
Brief Title: Indicators of Growth, Nutritional Status and Comorbide Disorders of Newborns With Down Syndrome
Acronym: DownSy
Status: Completed | Type: Observational
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Asija Rota Ceprnja, Asija Rota Ceprnja, MD., specialist of rehabilitation, University Hospital of Split
Other Study IDs: KBC2052018
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Down Syndrome,Auxological Indexes, Auxological Parametars, Intrauterine Growth Restriction
Keywords: growth restriction, nutritive status, comorbide disorders, Down Syndrome
MeSH Terms: conditions — Down Syndrome; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective To access predictive values of the auxological parameters and indexes for risk of comorbid malformations in newborns with Down syndrome (DS)

Study design In this cohort retrospective study, 141 newborns with proven trisomy 21 born at the Department of Gynecology and Obstetrics of the University of Split Hospital (1990 to 2015) were included. The data were obtained from the medical histories of mothers, infants and the delivery protocol.

The objective was to access predictive values of the auxological parameters and indexes for risk of comorbid malformations in newborns with Down syndrome (DS)

Conclusion Higher CI were found in hyportrophic (SGA) newborns with DS and indicated their intrauterine growth restriction with brain sparing and increased further risk of severe psychomotor retardation. The SGA newborns have lower parameters and indexes of nutritive status and significantly differed from eutrophic and hypertrophic newborns. These SGA newborns with DS have increased developmental risks and that requires further diagnostic attention.

DETAILED DESCRIPTION:
Use of anthropometric charts developed specifically for children with DS have a better expression of real growth restriction (small for gestation age/SGA, 9.9%) than the application of the percentile curve for typical children (SGA, 24.1%). These differences were also noted in the evaluation of other anthropometric measures. Cephalization index (CI) proved to be the only predictor from the considered auxological parameters and indexes with minimal predictive value in the prediction of heart defects type ASD II and VSD.

The presence of comorbid disorders in newborns with DS did not have a significant predictive role on growth indicators and nutritive status of the newborn, but we noted a strong association between preterm births and white matter injury (WMI).

ELIGIBILITY:
Inclusion Criteria:

The study included newborns with proven trisomy 21 born at the Department of Gynecology and Obstetrics of the University of Split Hospital Center from 1990 to 2015

Exclusion Criteria:

* excluded newborns with proven trisomy 21 died at first week of life

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The perinatal outcome of 141 children with confirmed diagnosis of DS was evaluated retrospectively. 137 (137/141, 97.2%) children had the cytogenetic finding of regular trisomy 21, 3 (3/141, 2.1%) had the kariotypic finding of mosaicism and 1 child (1/ 141. %) had translocation 21/22.
  There were more boys (74/141, 52.5%) than girls (67/141, 47.5%) in the examined sample.
  The median of gestational age of newborns with DS was 38 weeks (range 37-38 weeks): 10 children were born at 40 weeks of gestation (7.1%), 34 at 38 weeks (24.1%), 24 at 37 weeks (16.3%), 15 children (10.6%) at 36 weeks; and 19 children from 32 to 35 weeks of gestation.
  The median of gravidity for boys was the 3rd pregnancy, and for girls the 2nd pregnancy. The age range of the mother for both sexes was 31 to 35 years.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Categorization of subjects according to norms of growth rates for typical children and children with Down syndrome | 7 days
  Comparison of children with Down syndrome according to values of birth weight, birth length and head circumference classified by anthropometric charts for typical children and anthropometric charts for children with DS
Testing the differences of auxological characteristic according to gestational age | 7 days
  Comparison of auxological parameters and auxological indexes of premature and term babies with DS
Auxological characteristics of SGA, AGA and LGA children with DS by norms for DS | 7 days
  Comparison of auxological parameters and auxological indexes between hypotrophic (SGA), eutrophic (AGA) and hypertrophic (HGA) children with DS

CONTACTS AND LOCATIONS:
Overall Officials: Asija Rota Ceprnja, MD, Principal Investigator — University Hospital Split Department for Rehabilitation
Locations (1):
- Asija Rota Ceprnja, Split, Dalmatia, Croatia